CLINICAL TRIAL: NCT03316599
Title: Phase 1b Study of Gemcitabine, Nab-paclitaxel, and Ficlatuzumab (AV-299) in Patients With Advanced Pancreatic Cancer
Brief Title: Study of Gemcitabine, Nab-paclitaxel, and Ficlatuzumab (AV-299) in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Kimberly Perez, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-406
Record Dates: First submitted 2017-10-14; First posted 2017-10-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; ficlatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ficlatuzumab + Gemcitabine and Nab-Paclitaxel (Experimental): * Ficlatuzumab will be administered intravenously days 1 and 15 of a 28 day cycle
  * Gemcitabine 1000 mg/m2 and Nab-Paclitaxel 125mg/m2 will be administered IV days 1, 8, and 15 of a 28 day cycle.
  * Dosage of Ficlatuzumab is determined by dose level to which the patient is assigned at time of enrollment.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Ficlatuzumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Other Names: Gemzar
Drug: Nab-paclitaxel — Nab-paclitaxel is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells
  Other Names: Abraxane
Drug: Ficlatuzumab — It is selective recombinant humanized hepatocyte growth factor (HGF) inhibitory immunoglobulin G subclass 1 monoclonal antibody which blocks the MET tyrosine kinase receptor.

SUMMARY:
To identify the maximally tolerated dose of ficlatuzumab when combined with nab-paclitaxel and gemcitabine in patients with previously untreated pancreatic cancer.

DETAILED DESCRIPTION:
This research study is a Phase I dose-escalation clinical trial. It will test the safety and tolerability of an investigational drug ficlatuzumab when combined with Nab-paclitaxel and Gemcitabine, with the goal of determining the maximally tolerated dose of ficlatuzumab when combined with gemcitabine and nab-paclitaxel.

Ficlatuzumab is a type of drug called a "monoclonal antibody." It is thought to work by targeting hepatocyte growth factor (HGF) which is a HGF-c-Met inhibitor. The activation of the receptor tyroside kinase c-Met via its ligand, HGF, mediates proliferation, motility, and differentiation in a variety of cancers including pancreatic cancer.

Subjects must have a newly diagnosed stage 4 untreated metastatic pancreatic ductal cancer and meet all inclusion/exclusion criteria.

Treatment consists of 4 week treatment cycles. Ficlatuzumab will be administered on day 1 and 15 of each cycle. Nab-paclitaxel and gemcitabine will be administered on days 1,8, and 15.

Subjects continue in study until disease progression, adverse event/toxicity, death or either the subject or sponsor discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically- or histologically-confirmed pancreatic adenocarcinoma or poorly differentiated pancreatic carcinoma that is metastatic to distant sites.
* Other histologies such as neuroendocrine and acinar cell carcinoma are excluded.
* No prior chemotherapy for locally advanced or metastatic pancreatic cancer.
* Patients are eligible if they received adjuvant treatment after surgical resection with single-agent gemcitabine or gemcitabine/capecitabine or 5-fluorouracil/leucovorin that was completed >12 months before enrollment. Similarly, adjuvant radiation +/- chemosensitization with 5-fluorouracil, capecitabine, or gemcitabine is allowed if completed >12 months before enrollment.
* Participants are required to have measurable disease (RECIST v1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan. See section 11 for the evaluation of measurable disease.
* Participants enrolled must have disease that is accessible for tumor biopsies and must agree to a pre-treatment tumor biopsy.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (see Appendix A)
* Patients must have completed any major surgery or open biopsy ≥4 weeks from start of treatment.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤1.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Creatinine ≤1.5 × institutional upper limit of normal OR
  * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × upper limit of normal.
* Negative serum pregnancy test for women of childbearing potential.
* The effects of ficlatuzumab on the developing human fetus are unknown. For this reason and because Hepatocyte Growth Factor inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of ficlatuzumab administration.. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior chemotherapy or any other investigational agents for the treatment of locally advanced or metastatic pancreatic cancer
* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Screening for brain metastases with head imaging is not required.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ficlatuzumab or other agents used in study.
* History of prior or current synchronous malignancy, except:

  * Malignancy that was treated with curative intent and for which there has been no known active disease for >3 years prior to enrollment
  * Curatively treated non-melanoma skin cancer, cervical cancer in situ, or prostatic intraepithelial neoplasia, without evidence of prostate cancer
* Pre-existing, clinically significant peripheral neuropathy, defined as CTCAE grade 2 or higher neurosensory or neuromotor toxicity, regardless of etiology
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, NYHA class III/IV congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ficlatuzumab is hepatocyte growth factor inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ficlatuzumab, breastfeeding should be discontinued if the mother is treated with ficlatuzumab. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose of ficlatuzumab when administered in combination with gemcitabine and nab-paclitaxel | 2 years
  Identify maximally tolerated dose of ficlatuzumab when administered in combination with gemcitabine and nab-paclitaxel

SECONDARY OUTCOMES:
The response rate in this population of patients. | 2 years
  Determine the number of patients who demonstrate a clinical response assessed by RECIST criteria on imaging to the combination of ficlatuzumab with gemcitabine and nab-paclitaxel.
The progression free survival in this population of patients. | 2 years
  Determine the progression free survival derived from the combination of ficlatuzumab with gemcitabine and nab-paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No